CLINICAL TRIAL: NCT02615769
Title: Effect on Attendance if Including Focused Information of Spirometry in Preventive Health Checks - a Randomized Controlled Trial in Primary Health Care
Brief Title: Effect on Attendance if Including Focused Information of Spirometry in Preventive Health Checks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Randers Municipality, Denmark (Other); Central Denmark Region (Other); TRYG Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHPP-Lung
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2015-11

CONDITIONS: Spirometry; Patient Participation; Health Literacy; Lung Diseases
MeSH Terms: conditions — Patient Participation; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Invitation with focused information of spirometry (Experimental)
  Interventions: Behavioral: focused information of spirometry in the invitation
- Standard invitition (Active Comparator)
  Interventions: Behavioral: standard invitation

INTERVENTIONS:
Behavioral: focused information of spirometry in the invitation — Focused information of spirometry in the invitation to the preventive health check compose the intervention in this trial.
  Arms: Invitation with focused information of spirometry
Behavioral: standard invitation — The active comparator will receive a standard invitation to the preventive health checks. The preventive health checks in the active comparator group and the intervention group are identical.
  Arms: Standard invitition

SUMMARY:
The purpose of this study is to investigate if focused information of spirometry in the invitation to preventive health checks will increase the attendance compared with a standard invitation to preventive health checks.

DETAILED DESCRIPTION:
Background:

Lung diseases are among the most frequent and most serious ailments in Denmark. Chronic obstructive pulmonary disease (COPD) is the fourth most frequent cause of death and represents a significant burden on the health care system, the patients and their relatives. The National Board of Health in Denmark recommends spirometry to all individuals over 35 years who present at least one respiratory symptom (dyspnea, cough, wheeze or sputum production) or risk factors (prior or current smoking or relevant occupational exposure) in order to facilitate early detection of COPD. However approximately 200,000 citizens with COPD remain undiagnosed and unknown to the health care system.

Preventive health checks including spirometry can be used to detect lung diseases earlier. In a Danish municipality, the Check your Health Preventive Programme (CHPP) was initiated, offering preventive health checks to all 30 to 49 year-old citizens. This health promotion program provides the unique opportunity to evaluate single components of preventive health check in a real-life setting. Only a few previous studies have included spirometry in a preventive health check.

Over time the attendance at preventive health checks has decreased and at present the response rate is approximately 50%. Little is known about initiatives that can influence the attendance rate according to preventive health checks.

The aim of the study is to examine whether focused information on spirometry in the invitation material will influence the attendance in preventive health checks. The investigators hypothesize that spirometry as part of the preventive health check will increase the attendance in CHPP from 53% to 58% and the increase will be among prior and current smokers.

Materiel/Methods:

Check your health preventive program (CHPP):

The present study is embedded in the fourth year of the above mentioned CHPP. In CHPP, all citizens living in the municipality of Randers aged 30-49 years per 1st of January 2012 were identified in the Danish Civil Registration System. CHPP is a house-hold cluster randomized controlled trial offering a preventive health check to all 30 to 49 year old citizens in a Danish municipality during the years 2012 to 2017 (n= 26,216). The citizens were randomized by household into 5 groups of equal size, each corresponding to a specific year where they would be invited to a health check. Invitations with a prefixed appointment for the health check and information about the health check were dispatched continuously

Setting:

The health checks and the subsequent health behavioral courses are performed at a local health care center. The subsequent health interview takes place at the participants own general practitioner. The health checks will be conducted by health professionals who have experience with all measurement procedures as well as in risk communication to ensure standardization and quality.

The health check:

Prior to the health check the participants are asked to answer a web-based questionnaire regarding physical activity, self-rated health, mental health, smoking and alcohol. The clinical examination include following measures: biochemical (total cholesterol, lower density lipoprotein (LDL), glycated hemoglobin (HbA1c)), systolic and diastolic blood pressure, bodyweight, height, spirometry and Aastrands submaximal bike-test (cardiorespiratory fitness). At the end of the health check, the results are presented in a profile pamphlet including recommendations for follow up according to their risk-profile.

Execution of the health check is standardized by a written protocol and adherence is checked continuously.

Questionnaire:

Based on questionnaire data the following categorical variables will be described for all attendees:

* Age will be divided into four groups; 30-35, 36-40, 41-45 and 46-50
* Smoking status will be classified as smoker, ex-smoker, or never smoker and supplied with information about pack years.
* Airway symptoms (dyspnoea, wheezing or coughing) during the last four weeks will be divided into
* All of the time
* Most of the time
* Now and then
* Rarely
* Not at all

The present study:

This is a randomized controlled trial on attendance in preventive health check. From November 2015 until November 2016, 4,356 CHPP-citizens will be randomized further to either intervention or control in the present trial: The intervention group receives an invitation which highlights the value of spirometry as part of a health check. The invitation is made in collaboration with the Danish Lung Association and has been tested on a focus group before the invitations are dispatched. The control group will receive a standard invitation. Primary outcome measure is effect on attendance. Secondary outcome is the percentage of participants with abnormal spirometry assessed at the preventive health check. The characteristics of the 2 groups will be described according to sex, age, smoking history, spirometry values and lung symptoms. The intervention, the outcome and the group assignment in this trial are not revealed in the invitation for the citizens. Randomization is handled by an independent statistician.

Sample size:

The sample size is estimated to 4,356 participants in total and is calculated on the basis of the following assumptions: 1:1 randomization, two-sided significance level of 0.05, power of 0.9, intracluster correlation coefficient of 0.01 and with an average of 1.5 citizens in each household, we calculated the design effect to be 1.05. Calculations are further based on the objective of being able to detect a difference of 5% in effect size of attendance. The investigators determined this 5% difference to be clinically meaningful based on expert opinions and criteria employed in other research. The intracluster correlation coefficient was included to reflect a possible clustering effect of the general practitioners (n = 46), which is seldom greater than 0.01 in primary care settings.

Statistic analysis plan:

-The main outcomes Effect of the intervention on attendance will be estimated by differences in the proportion of citizens attending the health check in each of the groups. Crude and adjusted estimates of the difference in proportion will be based on binominal regression. Also these estimates will be compared with estimates based on propensity scores.

Furthermore, a descriptive analysis of attendees and non-attendees will be performed regarding sex, age, smoking history, self-reported lung symptoms and spirometry measurements. The analysis will follow the intention to treat principle.

For each of the endpoints, the number and percentage of individuals experiencing the endpoint will be presented, by randomisation group. Binominal regression will be used to estimate the difference in proportion between the two groups, and 95% confidence interval, comparing the intervention group with the comparison group. The baseline measure of the outcome will be included as a covariate in the model. If the distribution of the outcome is skewed, a log transformation will be used.

-Analysis of the baseline characteristics For the descriptive part of this study, bivariate and multivariate analysis will be performed. Continuous variables e.g. height and weight are presented as mean ± standard deviation, unless the variable has a highly skewed distribution, in which case, medians, 25th and 75th percentiles will be presented. For categorical variables, e.g. smoking status, civil status, and sex, the number and percentage of individuals within each category will be presented as absolute numbers and relative (%) frequencies. Anova will be used when comparing means or changes in means of numerical variables; and Chi2-test will be used when comparing proportions for categorical variables. Categorical outcomes will be analysed with logistic regression. The statistical significance level is set at p < 0.05. Statistical analysis will be performed using STATA 14.0 software.

Prevention of missing data :

The primary trial analysis will use an Intention To Treat (ITT) population, which includes all participants in the group to which they were randomised, regardless of the amount of intervention actually received. The only exclusion criterion is terminal illness as reported by the general practitioner.

To prevent attendees refusing to participate, households are invited together and two reminders are sent out. Furthermore, appointments are scheduled outside of work hours. Finally, we have the unique opportunity to use the Danish registers as a population-based health care database with information about the non-attendees, described below.

Treatment of missing data:

* Missing values due to incomplete clinical measurements or questionnaires Records with missing data due to incomplete questionnaires and incomplete spirometry measurements will be excluded. Sensitivity analysis will be performed and it will be considered if data are missing at random or not at random. Afterwards complete case analysis will be performed.
* Missing values of non-attendees As we have no clinical measurements or any answered questionnaires on the non-attendees, these data will be obtained from the Danish national registers. Sensitivity analysis will be performed and it will be considered if data are missing at random or not at random. Afterwards complete case analysis will be performed.
* Non-attendees will be described on following parameters:

  * Sociodemographic: Education level, sex, age, ethnicity and civil status from 2016 using Danish Civil Registration System(CRS)
  * Socioeconomics: income and transfer payments from 2016 using the Danish Civil Registration System(CRS) .
  * Contacts to their general practitioner from 2014-16 using reimbursement to the general practitioner from the Danish National Health Service Register.
  * Prescriptions of respiratory medicine from 2014-16 using the information about redeemed medication from the Danish National Prescription Register by using the ATC group R03 from 1995-2013. We categorized the drugs into rescue drugs against airway symptoms e.g. SABA / SAMA and chronic drugs against airway symptoms e.g. SABA/ SAMA, LABA/LAMA, leukotriene inhibitors, theophylline and inhaled corticosteroids.

Hypothesis:

The results from the present study are expected to contribute with important knowledge about the value of information on spirometry in invitations to health checks measured at different levels of attendance - as described above.

Legal and ethical aspects:

The study has been presented to The Scientific Ethics Committee and it is considered as routine data and thus ethical approval is not needed for the trial.

The study will comply with the declaration of Helsinki and according to the Danish Health Law each of the participants will provide written informed consent for data to be used for research. Approval by The Danish Data Protection Agency is obtained (2014-54-0704).

ELIGIBILITY:
Inclusion Criteria:

* Citizens in the municipality of Randers per 01.01.2012
* Randomized for the fourth group of five groups in total to be invited for a preventive health check as part of the health promotion program, Check your health prevention program, conducted in the years 2012 to 2017.

Exclusion Criteria:

* Terminal illness as reported by the citizens general practitioner.

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4496 (Actual)
Dates: Start 2015-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The percentage of participants attending the health check compared between the groups | one-year recruitment
  Primary outcome measure is effect of the focused information in the invitations on attendance.

SECONDARY OUTCOMES:
the percentage of participants with abnormal spirometry assessed at the preventive health | one-year recruitment
  Secondary outcome is the percentage of participants with abnormal spirometry assessed at the preventive health check.

CONTACTS AND LOCATIONS:
Overall Officials: Annelli Sandbæk, Professor, Study Chair — Institute of public health, section of general practice, Aarhus University
Locations (1):
- Institute of public health, section of general practice, Aarhus University, Aarhus C, Aarhus County, Denmark

REFERENCES:
- [Background] Adams G, Gulliford MC, Ukoumunne OC, Eldridge S, Chinn S, Campbell MJ. Patterns of intra-cluster correlation from primary care research to inform study design and analysis. J Clin Epidemiol. 2004 Aug;57(8):785-94. doi: 10.1016/j.jclinepi.2003.12.013. PMID 15485730
- [Background] Lauritzen T, Jensen MS, Thomsen JL, Christensen B, Engberg M. Health tests and health consultations reduced cardiovascular risk without psychological strain, increased healthcare utilization or increased costs. An overview of the results from a 5-year randomized trial in primary care. The Ebeltoft Health Promotion Project (EHPP). Scand J Public Health. 2008 Aug;36(6):650-61. doi: 10.1177/1403494807090165. PMID 18775821
- [Background] Hoj K, Skriver MV, Hansen AL, Christensen B, Maindal HT, Sandbaek A. Effect of including fitness testing in preventive health checks on cardiorespiratory fitness and motivation: study protocol of a randomized controlled trial. BMC Public Health. 2014 Oct 10;14:1057. doi: 10.1186/1471-2458-14-1057. PMID 25300392
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Fabricius P, Lokke A, Marott JL, Vestbo J, Lange P. Prevalence of COPD in Copenhagen. Respir Med. 2011 Mar;105(3):410-7. doi: 10.1016/j.rmed.2010.09.019. Epub 2010 Oct 16. PMID 20952174
- [Background] Riegels-Jakobsen T, Skouboe M, Dollerup J, Andersen CB, Staal LB, Jakobsen RB, Poulsen PB. Municipality screening of citizens with suspicion of chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2012;7:35-41. doi: 10.2147/COPD.S27314. Epub 2012 Feb 1. PMID 22315521
- [Background] Lokke A, Ulrik CS, Dahl R, Plauborg L, Dollerup J, Kristiansen LC, Cording PH, Dehlendorff C; TOP GOLD study-group. Detection of previously undiagnosed cases of COPD in a high-risk population identified in general practice. COPD. 2012 Aug;9(5):458-65. doi: 10.3109/15412555.2012.685118. Epub 2012 May 29. PMID 22643016
- [Background] Lauritzen T, Leboeuf-Yde C, Lunde IM, Nielsen KD. Ebeltoft project: baseline data from a five-year randomized, controlled, prospective health promotion study in a Danish population. Br J Gen Pract. 1995 Oct;45(399):542-7. PMID 7492424
- [Background] Lauritzen T, Nielsen KD, Leboeuf-Yde C, Lunde IM. [The health project Ebeltoft: health check ups and discussions in general practice. Basic data from a 5-year, prospective, randomized, controlled population study]. Ugeskr Laeger. 1997 Jun 16;159(25):3940-6. Danish. PMID 9214067
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; Consolidated Standards of Reporting Trials Group. CONSORT 2010 Explanation and Elaboration: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):e1-37. doi: 10.1016/j.jclinepi.2010.03.004. Epub 2010 Mar 25. PMID 20346624
- [Background] Lange P, Sondergaard J. [Early diagnosis of COPD is important and possible]. Ugeskr Laeger. 2013 Apr 29;175(18):1247-50. Danish. PMID 23651799
- [Background] Maindal HT, Stovring H, Sandbaek A. Effectiveness of the population-based Check your health preventive programme conducted in primary care with 4 years follow-up [the CORE trial]: study protocol for a randomised controlled trial. Trials. 2014 Aug 29;15:341. doi: 10.1186/1745-6215-15-341. PMID 25169211
- [Derived] Orts LM, Lokke A, Bjerregaard AL, Maindal HT, Norman K, Bech BH, Sandbaek A. The effect on participation rates of including focused spirometry information in a health check invitation: a cluster-randomised trial in Denmark. BMC Public Health. 2019 Aug 28;19(1):1183. doi: 10.1186/s12889-019-7531-5. PMID 31462261
- [Derived] Orts LM, Lokke A, Bjerregaard AL, Maindal HT, Sandbaek A. Effect on attendance by including focused information on spirometry in preventive health checks: study protocol for a randomized controlled trial. Trials. 2016 Dec 1;17(1):571. doi: 10.1186/s13063-016-1704-7. PMID 27906034
- See also: The Danish Lung Association — http://www.lunge.dk